CLINICAL TRIAL: NCT02630654
Title: Exploratory, Non-Interventional Study For Evaluating The Diagnostic, Prognostic And Response-Predictive Value Of A Multi Biomarker Approach In Metastatic GEP NETs
Brief Title: Study For Evaluating The Value Of A Multi Biomarker Approach In Metastatic GEP NETs
Acronym: EXPLAIN
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-99-52030-286
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen plasma will be saved in a biobank
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GEP NETs: Patients with a suspected diagnosis of metastatic GEP NETs
  Interventions: Other: This is a non-interventional study. Patients will be treated with any intervention deemed appropriate by the patient's physician.
- Healthy controls: Healthy controls matched by age and gender.
  Interventions: Other: This is a non-interventional study. Patients will be treated with any intervention deemed appropriate by the patient's physician.

INTERVENTIONS:
Other: This is a non-interventional study. Patients will be treated with any intervention deemed appropriate by the patient's physician.

SUMMARY:
This exploratory study aims to evaluate the diagnostic, prognostic and response predictive value of a multi biomarker strategy in patients with Gastroenteropancreatic Neuroendocrine Tumors (GEP NETs) originating from the midgut or pancreas. Using a recently developed methodology enabling the evaluation of 92 concomitant cancer biomarkers will provide an interesting approach to solve this question (Lundberg et al 2011).

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study related procedures.
* Suspected of suffering from a metastatic midgut NET or Pancreatic non-functional NET (WHO grade 1 or 2, up to 10% Ki67).
* Male or female aged 18 or older.

Exclusion Criteria:

* Previously treated for the NET disease with pharmaceutical treatment, Peptide Receptor Radionuclide Therapy (PRRT) or radiation therapy(surgery of primary tumour is accepted)
* Has any mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude.
* Suffering from a malignant disease or previously treated for a malignant disease within the last 6 months.
* Suffering from a chronic inflammatory disease.
* Suffering from a renal and/or liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from a specialist clinic with a suspected diagnosis of metastatic GEP NETs and healthy controls matched by age and gender.
Sampling Method: Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2014-03-24 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Progression Free Survival | Up to 60 months

SECONDARY OUTCOMES:
Change in oncological biomarker levels | Baseline visit and follow-up visit [i.e. every 3 months during the first year, every 6 months for the remainder of the study] up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (25):
- Denmark (3):
  - Aarhus
  - Copenhagen
  - Odense
- North Estonia Medical Center, Tallinn, Estonia
- Finland (3):
  - Helsinki
  - Oulu
  - Tampere
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East University Hospital, Riga
- Lithuania (4):
  - The Hospital of Lithuanian Health Science, Kaunas
  - Klaipėda University Hospital, Klaipėda
  - National Cancer Institute, Vilnius
  - Vilnius University Hospital, Vilnius
- Norway (4):
  - Bergen
  - Oslo
  - Stavanger
  - Trondheim
- Sweden (8):
  - Gothenburg
  - Jönköping
  - Lund
  - Örebro
  - Karolinska Universitetssjukhuset Bröst - och Endokrinkirurgiska kliniken, Stockholm
  - Södersjukhuset, Stockholm
  - Umeå
  - Uppsala

REFERENCES:
- [Derived] Kjellman M, Knigge U, Welin S, Thiis-Evensen E, Gronbaek H, Schalin-Jantti C, Sorbye H, Joergensen MT, Johanson V, Metso S, Waldum H, Soreide JA, Ebeling T, Lindberg F, Landerholm K, Wallin G, Salem F, Schneider MDP, Belusa R. A Plasma Protein Biomarker Strategy for Detection of Small Intestinal Neuroendocrine Tumors. Neuroendocrinology. 2021;111(9):840-849. doi: 10.1159/000510483. Epub 2020 Jul 28. PMID 32721955